CLINICAL TRIAL: NCT06965920
Title: Influence of Flexion Distraction Manipulation on Measures of Performance and Postural Control
Status: Enrolling by invitation | Type: Observational
Sponsor: Keiser University College of Chiropractic Medicine (Other)
Collaborators: Parker University (Other); Miami University (Other)
Responsible Party: Principal Investigator, Maruti Gudavalli, Professor, Keiser University College of Chiropractic Medicine
Other Study IDs: IRB000NV23MG145
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Spine Condition; Low Back Pain
Keywords: spine; low back pain; spinal manipulation; spinal mobilization; spinal stenosis
MeSH Terms: conditions — Low Back Pain; Spinal Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons receiving chiropractic care: Cox flexion distraction spinal manipulation/mobilization and other ancillary therapies as deemed fit by the treating clinician

SUMMARY:
This research study will evaluate human performance and postural balance changes during the course of care with flexion distraction manipulation in multiple chiropractic practices.

DETAILED DESCRIPTION:
Objective This research study will evaluate human performance and postural balance changes during the course of care with flexion distraction manipulation in multiple chiropractic practices.

Methods:

All patients who can stand without severe pain (able to stand normally at a 7 or below on qualitative analog visual pain scale [QVAS]) will be invited to participate. The goal is to recruit 150 participants from approximately 10 chiropractic practices. Volunteers will be given an informed consent document to read and if eligible and willing to participate will sign the informed consent document. At baseline and each subsequent testing visit, participants will complete the following:

* a numerical pain rating index (0-10) for each of the following: headache, neck pain, mid back pain and low back pain
* Keele STarT Back Screening Tool
* Assessment of Balance Confidence Questionnaire (ABC-6)
* Posture testing via force plate: Modified Test of Sensory Integration and Balance (MCTSIB), Single leg stance, limits of stability,
* Timed up and go and 5 times sit to stand tests The design of this study is observational, pre-post. Posture and performance testing is expected to last no more than 10 minutes per participant per visit. Subjective data will be captured via RedCap while objective data will be recorded by each clinician and uploaded to secure server.

The design of this study is observational, pre-post. Posture and performance testing is expected to last no more than 10 minutes per participant per visit. Subjective data will be captured via RedCap while objective data will be recorded by each clinician and uploaded to secure server.

ELIGIBILITY:
Inclusion Criteria:

* New patients with spinal pain,
* Patients will be between 18-100 years of age.
* All patients with spinal pain who - can safely stand and perform the basic parameters of the test at a 7 or below on qualitative visual analog scale (QVAS) on pain will be invited to participate.

Exclusion Criteria:

-Patients unable to stand normally with more than a 7 / 10 on the QVAS.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spinal pain presenting to participating Chiropractic clinics
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Modified Test of Sensory Integration and Balance (MCTSIB) score | From enrollment to end of 4 weeks and 8 weeks of treatment
  MCTSIB is a testing protocol available with BTracks balance system. Patients are asked to stand on a force plate for 20 seconds in four different conditions a) stand on a firm surface with eyes open b) stand on a firm surface with eyes closed c) stand on a foam with eyes open and d) stand on a foam with eyes closed. The path length of the center of pressure movement is quantified with a score. • Center of Pressure (COP) Path Lengths (PLs) under conditions of eyes open (EO), eyes closed (EC), eyes open foam (EOF), and eyes closed foam (ECF); higher values represent worse postural stability

SECONDARY OUTCOMES:
Numerical pain rating scale (0-10) on neck pain, mid-back pain, and low back pain | From enrollment to end of 4 weeks and 8 weeks of treatment
  Patients will enter the number corresponding to the level of pain in the three regions of the spine into a RedCap system. • Minimum value 0; Maximum value 10; higher values are worse pain scores
Limits of balance while standing on a force plate | From enrollment to end of 4 weeks and 8 weeks of treatment
  Patients will be asked to stand on a force plate and asked to lean forward, backward, and side ways (right and left). The limits of the center of pressure in anterior to posterior and lateral direction will be obtained using balance software. Center of pressure (COP) area is tested in four directions; front left (FL), back left (BL), back right (BR), and front right (FR) with an overall area provided; higher values represent better limits of stability
path length of center of pressure while standing on a single leg stance | From enrollment to end of 4 weeks and 8 weeks of treatment
  Patient will be asked to stand on a single leg for a maximum of 20 seconds. • Center of Pressure (COP) Path Lengths (PLs) for each leg and Asymmetry Index (ASI); higher COP values represent worse postural stability
Timed up and Go test in seconds | From enrollment to end of 4 weeks and 8 weeks of treatment
  Patients will be asked to get up from a chair and walk and time will be recorded. • Time in seconds to complete; greater time in seconds represents worse mobility and balance
time to Sit-to-stand test for 5 repetetions | From enrollment to end of 4 weeks and 8 weeks of treatment
  Patients will be asked to stand from a sitting position on a chair and repeated for 5 times. Time taken will be recorded.
  Time in seconds to complete; greater time in seconds represents worse lower extremity performance
• Keele STaRT Back | From enrollment to end of 4 weeks and 8 weeks of treatment
  The STarT Back Screening Tool helps primary care clinicians (GPs, physiotherapists etc) to group patients into three categories of risk of poor outcome (persistent disabling symptoms) - low, medium, and high-risk. By being able to categorise patients into these 3 groups, clinicians are then able to target interventions to each sub-group of patients to help outcome.
  Minimum value 0; Maximum value 9; higher values represent higher risk of poor outcome
• Assessment of Balance Confidence Questionnaire (ABC-6) | From enrollment to end of 4 weeks and 8 weeks of treatment
  This is a functional short form balance confidence questionnaire consisting of 6 questions with a scale of 0-100 for each question.
  Percent balance confidence - Minimum value 0%; Maximum value 100%; higher values represent greater balance confidence

CONTACTS AND LOCATIONS:
Overall Officials: Maruti R Gudavalli, PhD, Principal Investigator — Keiser University-West Palm Beach Campus; Ralph Kruse, DC, Study Director — Keiser University-West Palm Beach
Locations (1):
- Keiser University Spine care clinic, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will be shared as long as the receiving party signs confidentiality agreement